CLINICAL TRIAL: NCT06456320
Title: Mayo Clinic Tapestry 2.0: Applying Multi-Omics for Scientific Discovery
Status: Enrolling by invitation | Type: Observational
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Konstantinos N. Lazaridis, M.D., Executive Director, Center for Individualized Medicine, Mayo Clinic
Other Study IDs: 23-004120
Record Dates: First submitted 2024-06-07; First posted 2024-06-13 (Actual); Last update posted 2025-10-16 (Actual); Status verified 2025-09

CONDITIONS: Genetic Predisposition; Exposure, Environmental
MeSH Terms: conditions — Genetic Predisposition to Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Stool, urine, saliva, plasma, white blood cells (WBC), peripheral blood mononuclear cells (PBMC), whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Suspected Genetic Predisposition or Multi-Omics Contribution: Patients with a diagnosis or phenotype with the potential for association with a genetic predisposition or Multi-Omics Contribution.
- Healthy Control: Patients with no diagnosis associated with a genetic predisposition or Multi-Omics Contribution.

SUMMARY:
The purpose of this study is to use multi-omics testing on samples collected from Mayo Clinic patients to build and expand on what has been learned about genomic data.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Registered Mayo Clinic patient
* Able to provide informed written consent
* Able to receive mail and packages within a United States (US) state
* Able to collect and ship samples within a US state

Exclusion Criteria:

* Active hematological cancer or history of a hematological cancer
* Allogeneic Bone Marrow Transplant (e.g., samples from autologous bone marrow transplant recipients are acceptable if collected at least one month after transplant)
* Other co-morbidity that, in physician's opinion, would interfere with patient's ability to participate in the study (e.g., reduced ability to comprehend, i.e., dementia, intellectual disability, etc.)

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Mayo Clinic patients
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2024-09-05 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Creation of a unique integrated asset of multi-omics data | Up to 5 years
  A variety of patient cohorts will be ascertained throughout this study. Data will be made available to researchers to query correlations of disease states and clinical outcomes to multi-omics findings. These insights will be invaluable to creating omics-informed care plans in the future. Standard descriptive statistics approaches will be used for analysis.

CONTACTS AND LOCATIONS:
Overall Officials: Konstantinos N. Lazaridis, M.D., Principal Investigator — Mayo Clinic
Locations (3):
- United States (3):
  - Mayo Clinic in Arizona, Scottsdale, Arizona
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota

IPD SHARING:
Plan to Share IPD: Undecided